CLINICAL TRIAL: NCT00002664
Title: PHASE II STUDY OF MONOCLONAL ANTIBODY 17-1A WITH GM-CSF IN TREATMENT OF 5-FU RESISTANT COLORECTAL CANCER
Brief Title: Monoclonal Antibody Therapy and Colony- Stimulating Factor in Treating Patients With Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No recruitment
Sponsor: James Ahlgren (Other)
Responsible Party: Sponsor-Investigator, James Ahlgren, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWCC-5095; CDR0000064248 (Registry Identifier: PDQ (Physician Data Query)); NCI-V95-0686
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Edrecolomab; sargramostim

ARMS (1):
- Treatment (Experimental)
  Interventions: Biological: edrecolomab; Biological: sargramostim

INTERVENTIONS:
Biological: edrecolomab
Biological: sargramostim

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Colony-stimulating factors such as G-CSF may increase the number of immune cells found in bone marrow or peripheral blood, and may help a person's immune system kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of monoclonal antibody therapy plus G-CSF in treating patients with metastatic colorectal cancer that has not responded to treatment with fluorouracil.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response rate, duration of response, and survival after treatment with monoclonal antibody 17-1A and granulocyte-macrophage colony stimulating factor in patients with colorectal cancer metastatic to nonhepatic sites and refractory to fluorouracil. II. Describe the toxicities associated with this regimen. III. Assess the quality of life in these patients.

OUTLINE: Biological Response Modifier Therapy. Colorectal antigen 17-1A murine monoclonal antibody, MOAB 17-1A, NSC-377963; Granulocyte-macrophage colony stimulating factor (Immunex), GM-CSF, NSC-613795.

PROJECTED ACCRUAL: There will be 30 evaluable patients accrued into this study over approximately 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed carcinoma of the colon or rectum with radiologically confirmed metastases or clinically confirmed incurability No hepatic or CNS metastases Progression following fluorouracil (5-FU) alone or with a modulator (e.g., leucovorin, PALA, levamisole, interferon) Measurable disease outside prior radiotherapy fields The following are not considered measurable: Pleural effusion or ascites Osteoblastic lesions or evidence of disease on bone scan alone Progressive irradiated lesions alone Bone marrow involvement Brain metastases Malignant hepatomegaly by physical exam alone Chemical markers (e.g., CEA)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: At least 16 weeks Hematopoietic: Absolute neutrophil count at least 1,800/mm3 Platelet count at least 125,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Other: No concurrent infection Afebrile for at least 3 days prior to treatment unless fever due to tumor No known HIV infection No other medical condition that precludes protocol participation No second malignancy within 5 years except: Nonmelanomatous skin cancer Curatively treated in situ cervical carcinoma No pregnant or nursing women Negative pregnancy test required of fertile women Effective contraception required of fertile women Blood/body fluid analyses within 7 days prior to registration Imaging/exams for tumor measurement within 21 days prior to registration

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior mouse-based vaccines or monoclonal antibodies Chemotherapy: At least 2 weeks since prior 5-FU or at least 1 week past the AGC nadir, whichever is later No other prior chemotherapy except irinotecan Endocrine therapy: Not specified Radiotherapy: At least 6 months since radiotherapy Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1995-07; Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Ahlgren, MD, Study Chair — George Washington University
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States